CLINICAL TRIAL: NCT03431389
Title: "Outcomes of Tracheostomy Done for Patients Admitted in Anesthesia Intensive Care Units of Assiut University Hospital"
Acronym: PITS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor of anesthesia and intensive care, faculty of medicine, Assiut university., Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00008718/00045
Record Dates: First submitted 2018-02-03; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Tracheostomy Complication
MeSH Terms: interventions — Tracheostomy Decannulation

STUDY DESIGN:
Intervention Model Description: Tracheostomy done to all patients by open surgical technique and was done in ICUs without need to transfer to theatre. The patients were followed up daily until discharge from ICU. The following items were recorded: Duration of application of tracheostomy tube before decannulation (cannulation time), complications of tracheostomy, mortality due to tracheostomy.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decannulated group (Active Comparator): Decannulation was considered when the patients were no longer in need for tracheostomy tube and fulfilled the criteria of decannulation: No need for mechanical ventilation, no chocking with oral intake, no chest infection, effective cough reflex, laryngeal examination show bilateral mobile vocal cords with sufficient gap. Trial of decannulation was considered successful, if there was no need to reapply tracheostomy within 6 months of decannulation.
  Interventions: Device: Tracheostomy tube
- Failure of decannulation group (Active Comparator): Decannulation was considered when the patients were no longer in need for tracheostomy tube and fulfilled the criteria of decannulation: No need for mechanical ventilation, no chocking with oral intake, no chest infection, effective cough reflex, laryngeal examination show bilateral mobile vocal cords with sufficient gap. Decannulation trail was considered failed if there was a need to reapplication of tracheostomy at the time of decannulation or within six months of decannulation the duration of follow up.
  Interventions: Device: Tracheostomy tube

INTERVENTIONS:
Device: Tracheostomy tube — Tracheostomy done to all patients by open surgical technique and was done in ICUs without need to transfer to theatre.
  Other Names: TT

SUMMARY:
This study was undertaken to Identify the factors affecting the outcomes of tracheostomy done in ICU for patients subjected to prolonged intubation and ventilation and to suggest guidelines to control:

1. proper timing of tracheostomy
2. process of decannulation.

DETAILED DESCRIPTION:
Tracheostomy is described as the creation of a stoma at the skin surface which leads into the trachea. From the first tracheostomy until about 1930, the operation was performed exclusively for laryngeal obstruction. Nowadays, due to the development of the care of critically ill patients in intensive care units (ICUs), there are other indications for the procedure including prolonged intubation and pulmonary toilet.

The initial management of patients in an intensive care unit involves a series of interventions that aim to stabilize and then optimize their physiological state. Mechanical ventilation (MV) is a commonly utilized intervention to support a patient's respiratory function. The second phase in ICU management focuses on weaning the patient from the artificial supportive mechanisms.

The principle role of tracheostomy in the ICU is to expedite the weaning process in patients requiring prolonged mechanical ventilation and those predicted to be at risk of pulmonary aspiration. Tracheostomy facilitates weaning primarily by allowing increased level of patient activity and mobility.

Tracheostomy protects the larynx and the upper airway from prolonged intubation which may lead to laryngotracheal stenosis. Patients with tracheostomies tend to have fewer days of mechanical ventilation because of the improvements in the respiratory physiology. This is especially in trauma patients. They have improved secretion clearance as suction is easy and less strength is required for expectoration. This may be linked to the lower incidence of pneumonia and respiratory infections seen, especially in trauma victims.

Patients with tracheostomy are less sedated and therefore able to move in bed. The patients may also be able to swallow, so may be started on oral feeding sooner and mouth care is easier compared with an endotracheal tube (ETT) tube.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were admitted to the ICUs of the main Assiut University Hospital.
* mechanically ventilated and
* underwent tracheostomy during his/her stay in ICU.

Exclusion Criteria:

* Patients who were admitted to ICUs and didn't need tracheostomy during the period of admission in ICU or after discharge from ICU,
* Patients who died during admission in ICUs before being tracheostomized,
* Patients who died during admission in ICUs after being tracheostomized and the cause of death was not related to the tracheostomy procedure or care.

Ages: 1 Year to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Successful decanulation | 6 month
  Trial of decannulation was considered successful, if there was no need to reapply tracheostomy within 6 months of decannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor in anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt.
Locations (1):
- Assiut university main hospital, ICUs, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No